CLINICAL TRIAL: NCT02858310
Title: A Phase I/II Trial of T Cell Receptor Gene Therapy Targeting HPV-16 E7 for HPV-Associated Cancers
Brief Title: E7 TCR T Cells for Human Papillomavirus-Associated Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160154; 16-C-0154
Record Dates: First submitted 2016-08-04; First posted 2016-08-08 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09-02

CONDITIONS: Papillomavirus Infections; Cervical Intraepithelial Neoplasia; Carcinoma In Situ; Vulvar Neoplasms; Vulvar Diseases
Keywords: Immunotherapy; Human Papillomavirus; Vulvar Intraepithelial Neoplasia; Vulvar High Grade Squamous Intraepithelial Lesion; Vaccine; HPV-related Malignancy; HPV-related Carcinoma; HPV-related Cervical Carcinoma; HPV-related Anal Squamous Cell Carcinoma; HPV Positive Oropharyngeal Squamous Cell Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia; Carcinoma in Situ; Vulvar Neoplasms; Vulvar Diseases | interventions — aldesleukin; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Phase I (Experimental): Non-myeloablative, lymphocyte depleting preparative regimen, followed by E7 TCR Cells at escalating doses, followed by aldesleukin
  Interventions: Biological: E7 TCR cells; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide
- Arm 2: Phase II (Experimental): 1 x 10 e11 E7 Cells that was determined in Phase I + aldesleukin
  Interventions: Biological: E7 TCR cells; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: E7 TCR cells — T cells genetically engineered with a TCR targeting HPV-16 E7 (E7 TCR) that display specific reactivity against HLA-A2+, HPV-16+ target cells
Drug: Aldesleukin — Following cell infusion the patient receives high-dose bolus aldesleukin, which is dosed to individual patient tolerance. Aldesleukin improves the survival of E7 TCR cells after infusion.
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regimen.
Drug: Cyclophosphamide — Part of the non-myeloablative lymphocyte-depleting preparative regimen.

SUMMARY:
Background:

Human papillomavirus (HPV) can cause cervical, throat, anal, and genital cancers. Cancers caused by HPV have a HPV protein called E7 inside of their cells. In this new therapy, researchers take a person s blood, remove certain white blood cells, and insert genes that make them to target cancer cells that have the E7 protein. The genetically changed cells, called E7 TCR cells, are then given back to the person to fight the cancer. Researchers want to see if this can help people.

Objective:

To determine a safe dose and efficacy of E7 TCR cells and whether these cells can help patients.

Eligibility:

Adults ages 18 and older with an HPV-16-associated cancer, including cervical, vulvar, vaginal, penile, anal, or oropharyngeal.

Design:

Participants will list all their medicines.

Participants will have many screening tests, including imaging procedures, heart and lung tests, and lab tests. They will have a large catheter inserted into a vein.

Participants will have leukapheresis. Blood will be removed through a needle in the arm. A machine separates the white blood cells. The rest of the blood is returned through a needle in the other arm.

The cells will be changed in the lab.

Participants will stay in the hospital. Over several days, they will get:

Chemotherapy drugs

E7 TCR cells

Shots or injections to stimulate the cells

Participants will be monitored in the hospital up to 12 days. They will get support medicine and have blood and lab tests.

Participants will have a clinic visit about 40 days after cell infusion. They will have a physical exam, blood work, scans, and maybe x-rays.

Participants will have many follow-up visits with the same procedures. At some visits, they may undergo leukapheresis.

Participants will be followed for 15 years.

DETAILED DESCRIPTION:
Background:

* Metastatic or refractory/recurrent human papillomavirus (HPV)-16+ cancers (cervical, vulvar, vaginal, penile, anal, and oropharyngeal cancers) are incurable and poorly palliated by standard therapies.
* HPV-16+ cancers constitutively express the HPV-16 E7 oncoprotein, which is absent from healthy human tissues.
* Administration of T cell receptor (TCR) gene engineered T cells can induce objective tumor responses in certain malignancies including HPV-16+ cancers.
* T cells genetically engineered with a TCR targeting HPV-16 E7 (E7 TCR) display specific reactivity against HLA-A2+, HPV-16+ target cells.

Objectives:

Phase I Primary Objective

- To determine a safe dose for E7 TCR cells plus aldesleukin for the treatment of metastatic HPV-16+ cancers.

Phase II Primary Objective

-To determine safety and efficacy of E7 TCR cells plus aldesleukin for the treatment of metastatic HPV-16+ cancers.

Eligibility:

* Patients greater than or equal to 18 years old with metastatic or refractory/recurrent HPV-16+ cancer.
* Prior first line systemic therapy is required unless the patient declines standard treatment.
* Patients must be HLA-A*02:01-positive.

Design:

* This is a phase I/II clinical trial that will test the safety and efficacy of E7 TCR cells.
* All patients will receive a non-myeloablative lymphocyte-depleting preparative regimen of cyclophosphamide and fludarabine followed by a single infusion of E7 TCR cells. Cell infusion will be followed by high-dose aldesleukin.
* Re-enrollment will be allowed for a small number of subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic or refractory/recurrent HPV-16+ cancer (determined by in situ hybridization (ISH) or a polymerase chain reaction (PCR)-based test).
  2. Patients must be HLA-A*02 by low resolution typing, and HLA-A*02:01 by one of the high resolution type results.
  3. All patients must have received prior first line standard therapy or declined standard therapy.
  4. Patients with three or fewer brain metastases that have been treated with surgery or stereotactic radiosurgery are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for one month before protocol treatment. Patients with surgically resected brain metastases are eligible.
  5. Greater than or equal to 18 years of age.
  6. Able to understand and sign the Informed Consent Document.
  7. Clinical performance status of ECOG 0 or 1.
  8. Individuals must be willing to practice birth control from the time of enrollment on this study up to twelve (12) months after treatment. Individuals must be willing to undergo testing for HPV-16 prior to becoming pregnant after this period.
  9. Individuals of childbearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus. Individuals of childbearing potential are defined as all individuals except individuals who are postmenopausal or who have had a hysterectomy. Postmenopausal will be defined as individuals over the age of 55 who have not had a menstrual period in at least one year. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR transduced PBL, breastfeeding should be discontinued if the individual is treated with E7 TCR transduced PBL. These potential risks may also apply to other agents used in this study.
  10. Serology:
* Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
* Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.

  a. Hematology:
* Absolute neutrophil count greater than 1000/mm^3 without the support of

filgrastim.

* WBC greater than or equal to 3000/mm^3
* Platelet count greater than or equal to 100,000/mm^3
* Hemoglobin > 8.0 g/dL

  b. Chemistry:
* Serum ALT/AST less than or equal to 2.5 times the upper limit of normal
* Calculated creatinine clearance (CCr) greater than or equal to 50 mL/min/1.73^2 using the Cockcroft-Gault equation
* Total bilirubin less than or equal to 1.5 mg/dL, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dL

  c. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the E7 TCR cells.

Note: Patients may have undergone minor surgical procedures within the past three weeks, as long as all toxicities have recovered to Grade 1 or less.

EXCLUSION CRITERIA:

1. Active systemic infections (for e.g.: requiring anti-infective treatment), coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, severe obstructive or restrictive pulmonary disease. Patients with abnormal pulmonary function tests but stable obstructive or restrictive pulmonary disease may be eligible.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
4. Patients with autoimmune diseases such as Crohn s disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis or pancreatitis, and systemic lupus erythematosus. Hypothyroidism, vitiligo and other minor autoimmune disorders are not exclusionary.
5. Patients on immunosuppressive drugs including corticosteroids. With the exception of: intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)

   -Systemic corticosteroids at physiologic doses 10 mg/day of prednisone or equivalent;

   or,

   -Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
6. History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine or aldesleukin.
7. Patients with a history of coronary revascularization or ischemic symptoms unless patient has a normal cardiac stress test.
8. Documented LVEF of less than or equal to 45% tested. The following patients will undergo cardiac evaluations

   1. Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or
   2. Age greater than or equal to 50 years old
9. Any other condition, which would, in the opinion of the Principal Investigator, indicate that the subject is a poor candidate for the clinical trial or would jeopardize the subject or the integrity of the data obtained.
10. Subjects with baseline screening pulse oxygen level of < 95% on room air will not be eligible. If the underlying cause of hypoxia improves, then they may be reevaluated

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Phase II: Determine safety and effficacy of E7 TCR cells plus aldesleukin | At 12 weeks, every 3 months x 3, every 6 months x 5 years, then as per PI discretion thereafter
  Overall response rate (PR +CR)
Phase I: Determine a safe dose for E7 TCR cells plus aldesleukin | 30 days after treatment
  Number and type of AEs and/or UPs

SECONDARY OUTCOMES:
To assess progression-free survival | at time of last patient's progression
  time from start of treatment to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Draper LM, Kwong ML, Gros A, Stevanovic S, Tran E, Kerkar S, Raffeld M, Rosenberg SA, Hinrichs CS. Targeting of HPV-16+ Epithelial Cancer Cells by TCR Gene Engineered T Cells Directed against E6. Clin Cancer Res. 2015 Oct 1;21(19):4431-9. doi: 10.1158/1078-0432.CCR-14-3341. PMID 26429982
- [Background] Stevanovic S, Draper LM, Langhan MM, Campbell TE, Kwong ML, Wunderlich JR, Dudley ME, Yang JC, Sherry RM, Kammula US, Restifo NP, Rosenberg SA, Hinrichs CS. Complete regression of metastatic cervical cancer after treatment with human papillomavirus-targeted tumor-infiltrating T cells. J Clin Oncol. 2015 May 10;33(14):1543-50. doi: 10.1200/JCO.2014.58.9093. Epub 2015 Mar 30. PMID 25823737
- [Background] Hinrichs CS, Restifo NP. Reassessing target antigens for adoptive T-cell therapy. Nat Biotechnol. 2013 Nov;31(11):999-1008. doi: 10.1038/nbt.2725. Epub 2013 Oct 20. PMID 24142051
- [Derived] Nagarsheth NB, Norberg SM, Sinkoe AL, Adhikary S, Meyer TJ, Lack JB, Warner AC, Schweitzer C, Doran SL, Korrapati S, Stevanovic S, Trimble CL, Kanakry JA, Bagheri MH, Ferraro E, Astrow SH, Bot A, Faquin WC, Stroncek D, Gkitsas N, Highfill S, Hinrichs CS. TCR-engineered T cells targeting E7 for patients with metastatic HPV-associated epithelial cancers. Nat Med. 2021 Mar;27(3):419-425. doi: 10.1038/s41591-020-01225-1. Epub 2021 Feb 8. PMID 33558725
- [Derived] Jin BY, Campbell TE, Draper LM, Stevanovic S, Weissbrich B, Yu Z, Restifo NP, Rosenberg SA, Trimble CL, Hinrichs CS. Engineered T cells targeting E7 mediate regression of human papillomavirus cancers in a murine model. JCI Insight. 2018 Apr 19;3(8):e99488. doi: 10.1172/jci.insight.99488. eCollection 2018 Apr 19. PMID 29669936
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0154.html